CLINICAL TRIAL: NCT05791539
Title: Comparison Between Retrolaminar Block Combined With Erector Spinae Plane Block, and Erector Spinae Plane Block Alone for Post-thoracotomy Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, sherif Mamdouh Abbas, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MS-397-2022
Record Dates: First submitted 2022-12-16; First posted 2023-03-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Post-thoracotomy Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Randomization will be accomplished through the use of computer-generated random numbers and closed opaque envelopes. Another anesthesiologist who will not be involved in the other parts of the study will open the envelopes to enroll patients. and both patients and outcome assessors will be blinded to the assignment of groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 Erector spinae plane block (Experimental): Group 1 (ESPB (control group): (n = 15) patients will receive preoperative US-guided ESPB on the operated side by 20 ml bupivacaine 0.25%.
  Interventions: Procedure: Erector spinae plane block
- Group 2: Erector spinae plane block (Experimental): US-guided ESPB with 10 ml bupivacaine 0.25% (n = 15) on the operated side.
  Interventions: Procedure: Erector spinae plane block
- Retro laminar block (Experimental): the US-guided retrolaminar block 10 ml bupivacaine 0.25% group: (n = 15) on the operated side.
  Interventions: Procedure: erector spinae plane block + retrolaminar block

INTERVENTIONS:
Procedure: Erector spinae plane block — Patients will be divided into 2 groups group 1 will receive US-guided ESPB and group 2 will receive US-guided ESPB + US-guided Retrolaminar plain block before induction of GA.
  Arms: Group 1 Erector spinae plane block; Group 2: Erector spinae plane block
Procedure: erector spinae plane block + retrolaminar block — Patients will be divided into 2 groups group 1 will receive US-guided ESPB and group 2 will receive US-guided ESPB + US-guided Retrolaminar plain block before induction of GA.
  Arms: Retro laminar block

SUMMARY:
Post-thoracotomy pain is a challenging clinical problem that may be associated with increased morbidity and mortality. The current study tests two techniques of regional anaesthesia to control post thoracotomy pain

DETAILED DESCRIPTION:
Post-thoracotomy pain is a challenging clinical problem that may be associated with increased morbidity and mortality.

The surgical incision produces post-thoracotomy pain (PTP) via damage to the ribs and intercostal nerves, inflammation of the chest wall, pleura or pulmonary parenchyma cutting, and placement of the intercostal chest tube. Acute PTP inhibits the ability to breathe and cough normally. Numerous analgesic techniques are used to relieve PTP, including systemic opioids, regional techniques (such as paravertebral nerve blockade, intercostal nerve blockade, intrapleural analgesia, and epidural opioids with or without local analgesia), cryo-analgesia, and transcutaneous electrical nerve stimulation (TENS).

Emerging research has shown that the novel erector spinae plane block (ESPB) can be employed as a simple and safe alternative analgesic technique for acute post-surgical, post-traumatic, and chronic neuropathic thoracic pain in adults.

ESPB was first reported in 2016 for ipsilateral thoracic analgesia. It was found to be a safe and effective block that can be performed by an emergency physician in the emergency department setting for addressing acute pain due to multiple rib fractures.

Retrolaminar block (RLB) was first reported in 2006 as an alternative approach to PVB. RLB is performed with US imaging or the landmark technique. The efficacy of continuous RLB has been reported for breast cancer surgery .

However, the efficacy of ESPB has been described in a greater number of clinical reports than has RLB: a rib fracture, breast surgery, thoracoscopic surgery, lumbar spinal surgery, and laparoscopic abdominal surgery. In contrast to RLB, most of the literature on ESPB reported the use of the single-shot technique (80.2%). The local anesthetic was postulated to infiltrate the ventral and dorsal rami of the spinal nerve. However, Ueshima et al. reported that ESPB could not provide adequate analgesia of the anterior branch of the intercostal nerve.

The rationale of the study is that to the best of our knowledge each of ESPB and RLB has limitations regarding sensory block and distribution so our hypothesis is combining both will provide more solid block regarding sensory distribution, time interval of the block efficacy, and postoperative morphine consumption in patients undergoing thoracic surgeries.

Few studies evaluated the efficacy of ultrasound (US) guided erector spinae plane block on post-thoracotomy analgesia, however for the best of our knowledge no one compared the effect of ultrasound (US) guided retrolaminar block combined with erector spinae plane block and ultrasound (US) guided erector spinae plane block alone in patients undergoing thoracic surgeries.

ELIGIBILITY:
Inclusion Criteria:

* 1. Inclusion criteria

  * Age from 18-65 years.
  * body mass index (BMI) ranged between 20 and 40 kg/m2
  * ASA I, II patients undergoing open thoracic surgery through a posterolateral thoracotomy 2. Exclusion criteria
  * Patient refusal.
  * Sensitivity or contraindication to local anesthetic drugs.
  * History of psychological disorders and/or chronic pain.
  * Localized infection at the site of the block.
  * Coagulopathies, patients on anticoagulants and antiplatelets, and significant liver or renal insufficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-10-12 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Total amount of morphine consumption in the first 24-hour postoperative in the two groups. | 24 hours
  20ml for ESPB compared to 10ml ESPB added to 10ml RLB.

SECONDARY OUTCOMES:
•Pain score according to VAS score | 24 hours
  Pain score according to VAS score at 30min, 2h, 4h, 8h, 12h, 24h postoperative.
• Heart rate | intraoperative
  • Heart rate(Bpm) at 0 , 15min, 30min, 45min, 60min, 90min, 120min, then every 1h intraoperative.
Incidence of complications | 24 hours
  •Incidence of complications as hypotension, bradycardia, postoperative nausea, vomiting (PONV) and pruritis.
.First request of analgesia postoperative | 24 hours
  first time to request analgesia in the first 24 hrs
MAP | intraoperative
  Mean arterial blood pressure in mmhg at 0 , 15min, 30min, 45min, 60min, 90min, 120min, then every 1h intraoperative.

CONTACTS AND LOCATIONS:
Overall Officials: sherif mamdouh, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo Unviersity, Cairo, Egypt

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT05791539/Prot_SAP_000.pdf